CLINICAL TRIAL: NCT03603093
Title: Children's Hospital of Fudan University
Brief Title: A Multicenter Survey of the Indications for Esophagogastroduodenoscopy (EGD)
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Hunan Children's Hospital (Other Government); Wuhan Children's Hospital (Other); Xiamen Children's Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Other Study IDs: fudanU-E2
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Digestive System Abnormalities; Endoscopy
Keywords: Esophagogastroduodenoscopy; Paediatric
MeSH Terms: conditions — Digestive System Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Esophagogastroduodenoscopy (EGD) become more and more common in diagnosing gastroenterology diseases. The investigators want to find which symptoms can support for positive endoscopic findings through this multicenter study.

DETAILED DESCRIPTION:
Esophagogastroduodenoscopy (EGD) become more and more common in diagnosing gastroenterology diseases. And there are indications for EGD. Here, investigators want to find which symptoms can strongly support for positive endoscopy findings. So, investigators design the study to record the symptoms in detail and diagnosis, and then analysis symptoms and the rate of endoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients need esophagogastroduodenoscopic procedures

Exclusion Criteria:

* Patients whose parents reject to provide information for study

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All of the patients need esophagogastroduodenoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 2287 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Quantities of every indications for esophagogastroduodenoscopic procedures collected from questionaire finished by clinical doctor | from August 15th to October 15th in 2018
  Indications for esophagogastroduodenoscopic procedures were collected through questionaire, including abdominal pain, vomiting, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, doctor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan Universtity, Shanghai, China

REFERENCES:
- [Derived] Wang S, Qiu X, Chen J, Mei H, Yan H, You J, Huang Y. Pediatric esophagogastroduodenoscopy in china: indications, diagnostic yield, and factors associated with findings. BMC Pediatr. 2022 Sep 2;22(1):522. doi: 10.1186/s12887-022-03558-x. PMID 36056317